CLINICAL TRIAL: NCT01315158
Title: Incidence of Sedation Related Complications With Propofol Alone Versus Propofol With Benzodiazepines and Opiates in a High Risk Group Undergoing Advanced Endoscopic Procedures: A Randomized Controlled Trial
Brief Title: Propofol vs Propofol + Benzo/Opiates in High Risk Group
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: - The research team is not able to obtain the necessary support to continue the study.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-1133
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Sleep Apnea, Obstructive; Obesity
Keywords: Obstructive Sleep Apnea; Body Mass Index
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Propofol; Analgesics, Opioid; Benzodiazepines; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol+Benzo/Opioids (Active Comparator): If the patient is randomized into this arm the recommended Versed and Fentanyl doses are standardized:
  1. Recommended Versed:
     a. Prior to intubation
     * patient is < 50 kg = 1 mg Versed
     * patient is 50-75 kg = 1.5 mg Versed
     * patient is > 75 kg = 2 mg Versed
  2. Recommended Fentanyl
     1. Prior to intubation = 0.5 ug/kg
     2. Total procedural dose = 1 ug/kg
  Interventions: Drug: Propofol+Benzo/Opioids
- Propofol Alone (Active Comparator): The patients randomized into the sedation with propofol alone are able to cross over if they are unable to be successfully sedated under propofol alone. The the recommended doses before considering crossover are standardized:
  * Induction Dose: 2-2.5 mg/kg
  * Maintenance Dose: 0.1-0.2 mg/kg/min
  Interventions: Drug: Propofol Alone

INTERVENTIONS:
Drug: Propofol Alone — Recommended Propofol doses before considering crossover:
  * Induction: 2-2.5 mg/kg
  * Maintenance: 0.1-0.2 mg/kg/min
  Other Names: Propofol; Diprivan; 2,6-di-isopropofol
  Arms: Propofol Alone
Drug: Propofol+Benzo/Opioids — 1. Recommended Versed:
     a. Prior to intubation
     * patient is < 50 kg = 1 mg Versed
     * patient is 50-75 kg = 1.5 mg Versed
     * patient is > 75 kg = 2 mg Versed
  2. Recommended Fentanyl
     1. Prior to intubation = 0.5 ug/kg
     2. Total procedural dose = 1 ug/kg
  Other Names: Benzodiazepine; Midazolam; Versed; Opioid; Fentanyl
  Arms: Propofol+Benzo/Opioids

SUMMARY:
This will be a randomized controlled trial that compares the rates of sedation related complications in high risk patients (ASA greater or equal to 3, BMI greater or equal to 30, those at risk for OSA) undergoing advanced endoscopy procedures with propofol alone compared to propofol in combination with benzodiazepines and opioids.

DETAILED DESCRIPTION:
The use of propofol (2,6-di-isopropofol) for sedation during endoscopic procedures has increased in recent years primarily because of its favorable pharmacokinetic profile compared with traditional endoscopic sedation with benzodiazepines and opioids. Propofol has a rapid onset of action (30-45 sec) and short duration of effect (4-8 min). There also are data to support the safe use of propofol for advanced endoscopic procedures such as endoscopic retrograde cholangiopancreatography (ERCP) and endoscopic ultrasound (EUS).

There is limited information on the incidence of sedation related complications during advanced endoscopy. Prior studies were limited by controlled patient populations at low risk of developing sedation related cardiopulmonary complications. In a recent study, we defined the frequency of sedation related adverse events including the rate of airway modifications (AMs) with propofol use during advanced endoscopy. From a total of 799 patients, AMs were required in 14.4% of patients, hypoxemia in 12.8%, hypotension in 0.5% and premature termination in 0.6% of the patients. In addition, body mass index (BMI), male sex and American Society of Anesthesiologists (ASA) class of 3 or higher were independent predictors of AMs. Similarly, Wehrmann and Riphaus identified ASA class of 3 or higher, total propofol dose, history of alcohol use and having an emergency endoscopy as independent factors for sedation related complications in patients undergoing advanced procedures.

Given the alarming rates of obesity in the United States, it is believed that the prevalence of obstructive sleep apnea (OSA) may be 10% or higher and in obese adults these numbers could be as high as 25%. Using a previously validated screening tool for OSA [STOP-BANG (SB)], we reported a prevalence rate of patients at risk for OSA of 43.3% in patients undergoing advanced endoscopy procedures. Patients at risk for OSA with a positive SB score (score ≥ 3 of 8) had a higher rate of AMs (20% vs. 6.1%, adjusted relative risk 1.7) and frequency of hypoxemia (12% vs. 5.2%, adjusted relative risk 1.63) compared to those at low risk for OSA. Thus, based on the available data, it appears that ASA class 3 or higher, high BMI, and patients at risk for OSA are factors that place patients undergoing advanced endoscopy procedures at high risk for sedation related complications including airway modifications.

The optimal method for achieving deep sedation in this high risk group of patients is unclear. Propofol may accentuate airway collapse as patients become unresponsive to verbal stimulation (deep sedation). Recent studies suggest that propofol with midazolam and/or opioids may be synergistic in action and therefore the combined application of these drugs may permit smaller doses of each to be used and potentially lead to a reduction in risk of complications and in the dose of propofol needed while retaining the individual advantages of each compound. There is limited data evaluating the synergistic effect of propofol with midazolam and opioids in patients undergoing advanced endoscopy procedures. Ong and colleagues in a randomized controlled trial compared patient sedation and tolerance during ERCP using propofol alone or midazolam, ketamine and pentazocine (sedato-analgesic cocktail) for induction along with propofol for maintenance. Patient tolerance as assessed by visual analog scales by endoscopist and anesthetist were higher in the combination group. Paspatis et al reported higher dosage of intravenous propofol required in patients being sedated with propofol alone compared with that required in patients receiving oral dose of midazolam with propofol for ERCP procedures. In addition, the patients' anxiety levels before the procedure were lower in the combination group. The mean percentage decline in the oxygen saturation during the procedure was significantly greater in propofol alone group. However, these studies excluded patients deemed to be at a high risk for sedation related complications. Patients with ASA class 3 or higher were excluded, the mean BMI was less than 25, and included only patients at average risk for complications associated with sedation.

The significance of synergistic sedation in patients undergoing advanced endoscopy procedures in the high risk patients is unclear. The overall risk of sedation related complications is thought to be higher compared to standard endoscopy due to longer procedure times and the need for relatively deeper levels of sedation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Age greater than or equal to 18 years
* Presence of at least 1 of the following criteria:

  1. ASA class 3 or higher
  2. BMI of 30 or greater
  3. At risk for OSA (score of 3 or greater on the STOP-BANG screening tool)

Exclusion Criteria:

* drug allergy to Propofol, Benzodiazepines, or Opioids
* patients who received Benzodiazepines or Opioids within 24 hours of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faris Murad, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Rex DK, Deenadayalu VP, Eid E, Imperiale TF, Walker JA, Sandhu K, Clarke AC, Hillman LC, Horiuchi A, Cohen LB, Heuss LT, Peter S, Beglinger C, Sinnott JA, Welton T, Rofail M, Subei I, Sleven R, Jordan P, Goff J, Gerstenberger PD, Munnings H, Tagle M, Sipe BW, Wehrmann T, Di Palma JA, Occhipinti KE, Barbi E, Riphaus A, Amann ST, Tohda G, McClellan T, Thueson C, Morse J, Meah N. Endoscopist-directed administration of propofol: a worldwide safety experience. Gastroenterology. 2009 Oct;137(4):1229-37; quiz 1518-9. doi: 10.1053/j.gastro.2009.06.042. Epub 2009 Jun 21. PMID 19549528
- [Background] Standards of Practice Committee of the American Society for Gastrointestinal Endoscopy; Lichtenstein DR, Jagannath S, Baron TH, Anderson MA, Banerjee S, Dominitz JA, Fanelli RD, Gan SI, Harrison ME, Ikenberry SO, Shen B, Stewart L, Khan K, Vargo JJ. Sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2008 Nov;68(5):815-26. doi: 10.1016/j.gie.2008.09.029. No abstract available. PMID 18984096
- [Background] Tohda G, Higashi S, Wakahara S, Morikawa M, Sakumoto H, Kane T. Propofol sedation during endoscopic procedures: safe and effective administration by registered nurses supervised by endoscopists. Endoscopy. 2006 Apr;38(4):360-7. doi: 10.1055/s-2005-921192. PMID 16680635
- [Background] Rex DK, Heuss LT, Walker JA, Qi R. Trained registered nurses/endoscopy teams can administer propofol safely for endoscopy. Gastroenterology. 2005 Nov;129(5):1384-91. doi: 10.1053/j.gastro.2005.08.014. PMID 16285939
- [Background] Riphaus A, Stergiou N, Wehrmann T. Sedation with propofol for routine ERCP in high-risk octogenarians: a randomized, controlled study. Am J Gastroenterol. 2005 Sep;100(9):1957-63. doi: 10.1111/j.1572-0241.2005.41672.x. PMID 16128939
- [Background] Wehrmann T, Riphaus A. Sedation with propofol for interventional endoscopic procedures: a risk factor analysis. Scand J Gastroenterol. 2008 Mar;43(3):368-74. doi: 10.1080/00365520701679181. PMID 18938664
- [Background] Yusoff IF, Raymond G, Sahai AV. Endoscopist administered propofol for upper-GI EUS is safe and effective: a prospective study in 500 patients. Gastrointest Endosc. 2004 Sep;60(3):356-60. doi: 10.1016/s0016-5107(04)01711-0. PMID 15332023
- [Background] Vargo JJ, Zuccaro G Jr, Dumot JA, Shermock KM, Morrow JB, Conwell DL, Trolli PA, Maurer WG. Gastroenterologist-administered propofol versus meperidine and midazolam for advanced upper endoscopy: a prospective, randomized trial. Gastroenterology. 2002 Jul;123(1):8-16. doi: 10.1053/gast.2002.34232. PMID 12105827
- [Background] Paspatis GA, Manolaraki MM, Vardas E, Theodoropoulou A, Chlouverakis G. Deep sedation for endoscopic retrograde cholangiopancreatography: intravenous propofol alone versus intravenous propofol with oral midazolam premedication. Endoscopy. 2008 Apr;40(4):308-13. doi: 10.1055/s-2007-995346. Epub 2007 Dec 5. PMID 18058653
- [Background] Cote GA, Hovis RM, Ansstas MA, Waldbaum L, Azar RR, Early DS, Edmundowicz SA, Mullady DK, Jonnalagadda SS. Incidence of sedation-related complications with propofol use during advanced endoscopic procedures. Clin Gastroenterol Hepatol. 2010 Feb;8(2):137-42. doi: 10.1016/j.cgh.2009.07.008. Epub 2009 Jul 14. PMID 19607937
- [Background] Tishler PV, Larkin EK, Schluchter MD, Redline S. Incidence of sleep-disordered breathing in an urban adult population: the relative importance of risk factors in the development of sleep-disordered breathing. JAMA. 2003 May 7;289(17):2230-7. doi: 10.1001/jama.289.17.2230. PMID 12734134
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Hiestand DM, Britz P, Goldman M, Phillips B. Prevalence of symptoms and risk of sleep apnea in the US population: Results from the national sleep foundation sleep in America 2005 poll. Chest. 2006 Sep;130(3):780-6. doi: 10.1378/chest.130.3.780. PMID 16963675
- [Background] Cote GA, Hovis CE, Hovis RM, Waldbaum L, Early DS, Edmundowicz SA, Azar RR, Mullady DK, Jonnalagadda SS. A screening instrument for sleep apnea predicts airway maneuvers in patients undergoing advanced endoscopic procedures. Clin Gastroenterol Hepatol. 2010 Aug;8(8):660-665.e1. doi: 10.1016/j.cgh.2010.05.015. Epub 2010 May 23. PMID 20580942
- [Background] Cohen LB, Dubovsky AN, Aisenberg J, Miller KM. Propofol for endoscopic sedation: A protocol for safe and effective administration by the gastroenterologist. Gastrointest Endosc. 2003 Nov;58(5):725-32. doi: 10.1016/s0016-5107(03)02010-8. PMID 14595310
- [Background] Seifert H, Schmitt TH, Gultekin T, Caspary WF, Wehrmann T. Sedation with propofol plus midazolam versus propofol alone for interventional endoscopic procedures: a prospective, randomized study. Aliment Pharmacol Ther. 2000 Sep;14(9):1207-14. doi: 10.1046/j.1365-2036.2000.00787.x. PMID 10971238
- [Background] VanNatta ME, Rex DK. Propofol alone titrated to deep sedation versus propofol in combination with opioids and/or benzodiazepines and titrated to moderate sedation for colonoscopy. Am J Gastroenterol. 2006 Oct;101(10):2209-17. doi: 10.1111/j.1572-0241.2006.00760.x. PMID 17032185
- [Background] Reimann FM, Samson U, Derad I, Fuchs M, Schiefer B, Stange EF. Synergistic sedation with low-dose midazolam and propofol for colonoscopies. Endoscopy. 2000 Mar;32(3):239-44. doi: 10.1055/s-2000-134. PMID 10718390
- [Background] Cohen LB, Hightower CD, Wood DA, Miller KM, Aisenberg J. Moderate level sedation during endoscopy: a prospective study using low-dose propofol, meperidine/fentanyl, and midazolam. Gastrointest Endosc. 2004 Jun;59(7):795-803. doi: 10.1016/s0016-5107(04)00349-9. PMID 15173791
- [Background] Paspatis GA, Manolaraki M, Xirouchakis G, Papanikolaou N, Chlouverakis G, Gritzali A. Synergistic sedation with midazolam and propofol versus midazolam and pethidine in colonoscopies: a prospective, randomized study. Am J Gastroenterol. 2002 Aug;97(8):1963-7. doi: 10.1111/j.1572-0241.2002.05908.x. PMID 12190161
- [Background] Ong WC, Santosh D, Lakhtakia S, Reddy DN. A randomized controlled trial on use of propofol alone versus propofol with midazolam, ketamine, and pentazocine "sedato-analgesic cocktail" for sedation during ERCP. Endoscopy. 2007 Sep;39(9):807-12. doi: 10.1055/s-2007-966725. PMID 17703390
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Background] Aldrete JA, Kroulik D. A postanesthetic recovery score. Anesth Analg. 1970 Nov-Dec;49(6):924-34. No abstract available. PMID 5534693

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol+Benzo/Opioids: If the patient is randomized into this arm the recommended Versed and Fentanyl doses are standardized:
  1. Recommended Versed:
     a. Prior to intubation
     * patient is < 50 kg = 1 mg Versed
     * patient is 50-75 kg = 1.5 mg Versed
     * patient is > 75 kg = 2 mg Versed
  2. Recommended Fentanyl
     1. Prior to intubation = 0.5 ug/kg
     2. Total procedural dose = 1 ug/kg
  Propofol+Benzo/Opioids: 1. Recommended Versed:
  a. Prior to intubation
  * patient is < 50 kg = 1 mg Versed
  * patient is 50-75 kg = 1.5 mg Versed
  * patient is > 75 kg = 2 mg Versed
    2. Recommended Fentanyl
    a. Prior to intubation = 0.5 ug/kg b. Total procedural dose = 1 ug/kg
- Propofol Alone: The patients randomized into the sedation with propofol alone are able to cross over if they are unable to be successfully sedated under propofol alone. The the recommended doses before considering crossover are standardized:
  * Induction Dose: 2-2.5 mg/kg
  * Maintenance Dose: 0.1-0.2 mg/kg/min
  Propofol Alone: Recommended Propofol doses before considering crossover:
  * Induction: 2-2.5 mg/kg
  * Maintenance: 0.1-0.2 mg/kg/min
Period: Overall Study
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Started | 17 | 19
Completed | 17 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 8 | 14 | 22
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience Airway Maneuvers
Description: In high risk patients (meeting at least of 1 of 3 criteria: ASA ≥ 3, BMI ≥ 30, those at risk for OSA) undergoing advanced endoscopy procedures, compare the number of participants who experience airway maneuvers (AMs) when sedated with propofol alone versus propofol in combination with benzodiazepines and opioids.
Time Frame: One day (during procedure)
Measure: Number; unit: participants
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Number analyzed (Participants) | 17 | 19
participants | 4 | 4

2. Secondary Outcome: Number of Participants Who Experience Other Sedation Related Complications
Description: Compare the number of participants who experience other sedation related complications such as hypotension, hypoxemia and need for termination of the procedure between the two groups
Time Frame: One day (during procedure)
Measure: Number; unit: participants
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Number analyzed (Participants) | 17 | 19
participants | 0 | 0

3. Secondary Outcome: Compare Propofol Doses Between the Two Groups
Description: The dose of propofol used between the two groups will be compared
Time Frame: One day (during procedure)
Population: The data for this outcome measure was not collected and was not analyzed due to not having the necessary support to continue the study.
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Predictors of Sedation Related Complications as Measured by the Number of Participants Who Experience Hypoxemia (Defined as a Pulse Oximetry <90% for Any Duration)
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Number analyzed (Participants) | 17 | 19
participants | 0 | 0

5. Secondary Outcome: Predictors of Sedation Related Complications as Measured by Hypopnea/Apnea (Defined as Fewer Than 6 Breaths/Minute Based on Capnography)
Time Frame: One year
Measure: Number; unit: incidences
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Number analyzed (Participants) | 17 | 19
incidences | 0 | 0

6. Secondary Outcome: Predictors of Sedation Related Complications as Measured by the Incidences of Hypotension (Defined as Systolic Blood Pressure of Less Than 90mmHg or a Decrease of More Than 25% From Baseline)
Time Frame: One year
Measure: Number; unit: incidences
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Number analyzed (Participants) | 17 | 19
incidences | 0 | 0

7. Secondary Outcome: Predictors of Sedation Related Complications as Measured by Early Procedure Termination for an Alternative Sedation Related Complication
Time Frame: One year
Measure: Number; unit: incidences
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Number analyzed (Participants) | 17 | 19
incidences | 0 | 0

8. Secondary Outcome: Patient Tolerance as Assessed by Endoscopists
Description: The frequency of symptoms of nausea and vomiting in the two groups of patients will be recorded. Patient tolerance of the procedure will be assessed independently by the endoscopist using a 100-mm visual analog scale (VAS, 0=unmanageable, 100=excellent). The patient will also score the level of tolerance using the same VAS at a routine follow-up phone call made 24-48 hours after the procedure.
Time Frame: 24-48 hours
Population: as for outcome 3
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants Who Experience Symptoms of Nausea and Vomiting Will be Compared Between the Two Groups
Description: The number of participants who experience symptoms of nausea and vomiting in the two groups of patients will be recorded. This will be recorded during the follow-up phone call made 24-48 hours after the procedure.
Time Frame: 24-48 hours
Measure: Number; unit: participants
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Number analyzed (Participants) | 17 | 19
participants | 2 | 1

ADVERSE EVENTS:
Arm/Group | Propofol+Benzo/Opioids | Propofol Alone
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes